CLINICAL TRIAL: NCT02808728
Title: Effectiveness of Intraoperative Exparel, a Bupivacaine Liposome Injectable Suspension, for Postoperative Pain Control in Total Knee Arthroplasty: A Prospective, Randomized, Double Blind, Controlled Study
Brief Title: Effectiveness of Intraoperative Exparel for Postoperative Pain Control in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: DeClaire LaMacchia Orthopaedic Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WIRB 20131914
Record Dates: First submitted 2016-06-14; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis; Total Knee Arthroplasty; Pain Management
Keywords: Total Knee Arthroplasty; Total Knee Replacement; Exparel; Liposomal Bupivacaine; Ropivacaine; Postoperative Pain Management
MeSH Terms: conditions — Osteoarthritis; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pain Cocktail with Ropivacaine (Active Comparator): patients given the standard intra-articular "pain cocktail" injection, consisting of ropivacaine, ketorolac, morphine, and epinephrine mixed with saline into a 100cc preparation.
  given in one single dose
  Interventions: Drug: Pain Cocktail with Ropivacaine
- Pain Cocktail with Exparel (Experimental): patients given a similar intra-articular injection consisting of bupivacaine, ketorolac, morphine, and epinephrine mixed with saline into a 80cc preparation as well as an injection of Exparel, 20cc of 1.3% Exparel, to total 100cc.
  given in one single dose
  Interventions: Drug: Pain Cocktail with Exparel

INTERVENTIONS:
Drug: Pain Cocktail with Exparel — pain cocktail: bupivacaine, ketorolac, morphine, and epinephrine mixed with saline into a 80cc preparation as well as an injection of Exparel (bupivacaine liposome injectable suspension), 20cc of 1.3% Exparel, to total 100cc.
  Other Names: liposomal bupivacaine
  Arms: Pain Cocktail with Exparel
Drug: Pain Cocktail with Ropivacaine — pain cocktail: ropivacaine, ketorolac, morphine, and epinephrine mixed with saline into a 100cc preparation.
  Arms: Pain Cocktail with Ropivacaine

SUMMARY:
Does the use of periarticular Exparel in total knee arthroplasty prove to more effectively manage post operative pain control than another local analgesic, Ropivacaine, when both are used as part of a multimodal pain management approach?

The investigators hypothesize that Exparel, a bupivacaine liposomal injectable suspension, will improve total knee arthroplasty postoperative pain with significant improvement of early function outcomes.

DETAILED DESCRIPTION:
The investigators use a double blind, controlled, randomized study to examine the effectiveness of periarticular Exparel in total knee arthroplasty postoperative pain control as well as effect on early mobilization and length of hospital stay when compared to another local analgesic (Ropivacaine) when both are used as part of a multimodal pain management approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing Total Knee Arthroplasty with Dr. J.H. DeClaire
* 18 years of age or older
* Primary diagnosis of osteoarthritis of the knee
* Opioid naïve patient (according to FDA guidelines)

Exclusion Criteria:

* Prior knee replacement
* Prior use of narcotics for chronic pain management
* Inflammatory arthritis (Rheumatoid arthritis, Lupus, etc.)
* Unicompartmental knee replacement
* Bilateral Total Knee Arthroplasty
* Opioid Tolerant as defined by the FDA: Patients who are taking, for one week or longer, at least:

> 60 mg oral morphine/day > 25μg transdermal fentanyl/hour > 30 mg oral oxycodone/day > 8 mg oral hydromorphone/day > 25 mg oral oxymorphone/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid consumption | immediately post-operatively through hospital stay
  oral and intravenous narcotic consumption is recorded during hospital stay

SECONDARY OUTCOMES:
Hours to ambulate 100 feet | immediately post-operatively through hospital stay
Length of hospital stay (hours) | immediately post-operatively through hospital stay
  Number of hours the patient stays at the hospital following operation
Visual Analog Pain Score | day 1 and day 2 after operation, 3 months, 6 months, and 1 year operatively
Knee Society Score | 3 months, 6 months, 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Olayinka Warritay, MD, Study Director — DeClaire LaMacchia Orthopaedic Institute

REFERENCES:
- [Derived] DeClaire JH, Aiello PM, Warritay OK, Freeman DC. Effectiveness of Bupivacaine Liposome Injectable Suspension for Postoperative Pain Control in Total Knee Arthroplasty: A Prospective, Randomized, Double Blind, Controlled Study. J Arthroplasty. 2017 Sep;32(9S):S268-S271. doi: 10.1016/j.arth.2017.03.062. Epub 2017 Apr 6. PMID 28478185